CLINICAL TRIAL: NCT05013801
Title: A Randomized, Controlled, Single Center Clinical Study to Evaluate the Effect of Facial Serum Q69 in Moderating the Appearance of Mild to Moderate Melasma
Brief Title: A Clinical Study to Evaluate the Effect of Facial Serum Q69 in Moderating the Appearance of Mild to Moderate Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Shanghai Skin Disease and Venereal Disease Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKN-SFF-3469
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Melasma
Keywords: face
MeSH Terms: conditions — Melanosis; Facies | interventions — hydroquinone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cosmetic Facial Serum Q69 (Experimental): Cosmetic facial serum. To be used twice daily on lesional areas of the face for 12 weeks.
  Interventions: Other: Cosmetic facial serum Q69
- 2% Hydroquinone (Other): 2% hydroquinone cream to be used twice daily on lesional areas of the face as directed by the dermatologist for no longer than 8 weeks.
  Interventions: Drug: 2% Hydroquinone

INTERVENTIONS:
Other: Cosmetic facial serum Q69 — Cosmetic facial serum
  Arms: Cosmetic Facial Serum Q69
Drug: 2% Hydroquinone — 2% Hydroquinone cream
  Arms: 2% Hydroquinone

SUMMARY:
This is a single centre, 2-cell, single blinded full-face (products applied at lesional sites) study to evaluate changes in melasma through a cosmetic facial serum formulation and marketed 2% Hydroquinone product

DETAILED DESCRIPTION:
This is a single blind (outcomes assessor), randomized, 2 cell, full face study to evaluate changes in mild malar melasma through use of a cosmetic facial serum formulation or marketed 2% hydroquinone. This study will accept up to fifty participants per cell (100 participants overall) who meet the inclusion/exclusion criteria to ensure that at least forty participants per cell complete the study. Participants will be randomized to receive either the cosmetic product or the hydroquinone product.

The study schedule will be different depending which product the subject is allocated to.

If accepted onto the study, all participants will be provided with a marketed face wash and moisturiser to use for one week before the baseline visit.

At the baseline visit, following collection of baseline measures subjects will be allocated to either the cosmetic product or 2% hydroquinone. Products will be applied only to lesional areas on the face twice daily. Participants will also be provided with a sunscreen for use throughout the test phase of the study. They will continue to use the face wash and moisturiser with which they have previously been provided.

Participants allocated to the cosmetic product will be asked to return to the study centre for assessments at weeks 4, 8, 12 and regression (8 weeks after stopping product application).

Participants allocated to 2% hydroquinone will be asked to return to the study centre 3 days, 1, 2, 4, 6 and 8 weeks after baseline and regression 8 weeks after stopping product application).

ELIGIBILITY:
Inclusion Criteria:

* Participant in general good health as per the Medical History screening criteria
* Female participants between 18-55 years of age at first study visit (both inclusive)
* Participant having mild to moderate facial melasma
* Participants having skin type II-IV
* Participants with melasma pigmentation which has been stable for 3 months (self-reported)
* Participants who are willing to dedicate time and follow the instructions as per the study protocol
* Participants willing to give a voluntary written informed consent for activities in the study for imaging and agree to come for regular study visits

Exclusion Criteria:

* Participants are pregnant or anticipating pregnancy during the study period or are currently breast-feeding as self-reported
* Participants with known allergies to facial skin care products including sunscreens, bar or liquid cleansing products, moisturizers/lotions, lightening/brightening products, antiaging products, adhesives, and/or fragrances
* Participants who are consistently exposed to sunlight either through their work or habits, such as continuous exposure to sunlight that is more than 2 hours of duration.
* Participants who have sunburn, suntan, scars, nevi, excessive hair, tattoos, birthmarks, or any other dermal conditions on the test sites that might influence the test results in the opinion of the Investigator
* Participant with dry or scaly facial skin or with self-perceived pimple prone &/or sensitive skin or with any other signs of significant local irritation
* Participants having a history or currently having skin conditions such as eczema or psoriasis, severe acne, nodules, cyst, eczema, seborrheic dermatitis, severe excoriations on the face currently or in adult life
* Participants allergic to sulphite containing drugs
* Participants who have used any medication (including Hydroquinone, retinoids) in the last two 2 months for melasma treatment
* Participants not tolerant to retinoids or Vitamin-A related medicines or products
* Participants with a history of Asthma, Hypertension, diabetes, or any other illness that the Investigator deems inappropriate for participation or could interfere with the study outcome
* Participants taking medication continuously/regularly every day such as corticosteroids or non-steroidal anti-inflammatories, topically for four weeks or orally for eight weeks prior to the study
* Participants who are currently participating in any clinical study
* Participants who have participated in any clinical trial involving the face in the past 8 weeks prior to inclusion into this study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Change in L* | 0 - 12 weeks + regression (8 weeks)
  CIELAB colour space L* (perceptual lightness), measured using Konica Minolta CM-2600d portable spectrophotometer
Change in modified Melasma Area Severity Index (mMASI) | 0 - 12 weeks + regression (8 weeks)
  Melasma severity on four facial areas (forehead, right malar region, left malar region and chin) is assessed based on three variables: percentage of the total area involved (A), darkness (D), and homogeneity (H).
  Area (A): a numerical value is assigned to % area involved as follows. 0=no involvement; 1=<10% ; 2=10-29%; 3=30-49%; 4=50-69%; 5=70-89%; and 6=90-100%.
  Darkness of melasma (D) is graded on a scale of 0 to 4: 0=normal skin color without evidence of hyperpigmentation; 1=barely visible hyperpigmentation; 2=mild hyperpigmentation; 3=moderate hyperpigmentation; 4=severe hyperpigmentation.
  Homogeneity of hyperpigmentation (H) is graded on a scale of 0 to 4 as follows: 0=normal skin color without evidence of hyperpigmentation; 1=specks; 2=small patchy areas <1.5 cm diameter; 3= >2 cm diameter; 4=uniform skin involvement without any clear areas.
  The sum of D and H is multiplied by A and by the percentages of the four facial areas (10-30%).
  Total score is 0-48.

SECONDARY OUTCOMES:
Change in evenness of skin tone | 0 - 12 weeks + regression (8 weeks)
  Evenness of skin tone as assessed through analysis of images captured using the Canfield Scientific VISIA-CR imaging system
Change in visual skin glow | 0 - 12 weeks + regression (8 weeks)
  Composite parameter calculated using output from CM2600d and VISIA-CR

OTHER OUTCOMES:
Change in perception of melasma as assessed using MelasQOL | 0 - 12 weeks + regression (8 weeks)
  Quality of life questionnaire specifically developed for use with melasma

CONTACTS AND LOCATIONS:
Overall Officials: Yimei Tan, MD, Principal Investigator — Shanghai Skin Disease Hospital
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No